CLINICAL TRIAL: NCT05401617
Title: Impact of an Information Assistance Application in Addition to a Traditional Anesthesia Consultation on Preoperative Anxiety in Pediatrics: Prospective Randomized Trial
Acronym: Anx'Appli
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2019/0087/HP
Record Dates: First submitted 2022-05-20; First posted 2022-06-02 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Pediatric Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): patient benefiting from a traditional anesthesia consultation as performed daily in the department (control group). The information will be delivered according to local customs and the MAR: oral, which can be supplemented by the delivery of the SPARADRAP booklet and the written documents usually delivered
- experimental group (Experimental): patient benefiting, in addition to this traditional anesthesia consultation, from additional information via the computerized tool. The operation of this tool will be explained by paramedical staff and its access will be free as soon as you leave the consultation.
  Interventions: Other: additional information via the computerized tool

INTERVENTIONS:
Other: additional information via the computerized tool — additional information delivered via the computerized tool
  Arms: experimental group

SUMMARY:
The objective of the study is to evaluate the benefits on pre-operative anxiety of an information assistance application in addition to a traditional anesthesia consultation on preoperative anxiety in pediatrics

ELIGIBILITY:
Inclusion Criteria:

* Child between 4 years old (inclusive) and 10 years old (inclusive);
* Must benefit from programmed general anesthesia for scheduled surgery at the Rouen University Hospital, in the paediatrics ward;
* Benefiting from a social security scheme;
* Whose parental authority has consented to participation in the research;
* Not having expressed their refusal to participate in the research;
* Understanding French;
* Ability to access the application being researched.

Exclusion Criteria:

* Patient with cognitive disorders: disorders known in the history and assessed or suspected during the anesthesia consultation.
* Poor understanding of oral French by the child;
* Poor understanding of the oral and/or written French language by the parent/legal representative;
* Patient presenting a contraindication to general anesthesia or to the intervention during the pre-anaesthetic visit;
* Patient with severe psychiatric disorders

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 182 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Level of anxiety on entering the operating room | 15 days
  YALE score (also called m-YPAS SF) : 22.9 to 100

SECONDARY OUTCOMES:
Anxiety of parents | 15 days
  EVA (Analogic Visual Scale) score : 0 to 10
Need of an analgesic supplement in SSPI (post-interventional monitoring room) | 15 days
Duration of stay in SSPI | 15 days
  Stay in SSPI in minutes
Parents' satisfaction with the quality of the information provided | 15 days
  numerical scale : 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Compere, Principal Investigator — University Hospital, Rouen
Locations (1):
- UHRouen, Rouen, France